CLINICAL TRIAL: NCT01055782
Title: Kan Anvendelse af Endoskopisk Positioneringsudstyr Ved coloskopiundersøgelsen (kikkertundersøgelse af Tarmen) i en højt Specialiseret Praksis Forbedre Patientens Subjektive Kvalitetsoplevelse (Smerteperception)?
Brief Title: Colonoscopy Endoguide in Specialist Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Specialist Doctors at Rolighedsvej (Other)
Collaborators: Danish Medical Association (Other); Surgical Clinic, Allerød, Denmark (Unknown)
Responsible Party: Principal Investigator, Lene Hendel, MD, DMsc, The Specialist Doctors at Rolighedsvej
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-1-2009-80
Record Dates: First submitted 2010-01-24; First posted 2010-01-26 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Colonoscopy; Pain
Keywords: Colonoscopy; Endoguide; Pain perception; Colonoscopy to the coecum (success rate); Patient's perception of pain; Duration of successful colonoscopies
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With endoguide (Experimental): Colonoscopy completed with endoguide
  Interventions: Device: Endoguide
- Without endoguide (No Intervention): Colonoscopy completed without endoguide

INTERVENTIONS:
Device: Endoguide — Use of endoguide to facilitate completion of endoscopy
  Arms: With endoguide

SUMMARY:
The study includes 700 patients referred for colonoscopy are randomized to colonoscopy with or without endoguide.

The study will investigate whether the endoguide improves success rate and the patient's perception of pain.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent provided

Exclusion Criteria:

* Informed consent not provided or not possible to obtain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1004 (Actual)
Dates: Start 2009-11; Primary Completion 2011-04 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Speciallægerne på Rolighedsvej, Birkerød, Birkerød, Denmark

REFERENCES:
- [Derived] Bak-Christensen A, Knudsen E, Hendel J, Ifaoui IB, Lehrskov-Schmidt L, Hendel L. Colonoscopy results are not enhanced by use of magnet endoguide in specialist practice. Dan Med J. 2013 Jun;60(6):A4611. PMID 23743108

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | With Endoguide | Without Endoguide
Started | 555 | 449
Completed | 555 | 449
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | With Endoguide | Without Endoguide | Total
Number analyzed (Participants) | 555 | 449 | 1004
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 382 | 297 | 679
  >=65 years | 173 | 152 | 325
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (14) | 56 (15) | 56 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 308 | 256 | 564
  Male | 247 | 193 | 440
Region of Enrollment [Number; unit: participants]
  Denmark | 555 | 449 | 1004

OUTCOME MEASURES:

1. Primary Outcome: Completed Colonoscopy
Time Frame: immediately after colonoscopy
Population: Choosen by randomization.
Measure: Number; unit: participants
Groups:
- With Endoguide - Success Rate: Exams completed with endoguide. Success rate/completion.
- Without Endoguide: Exams completed without endoguide. Success rate/completion.
Arm/Group | With Endoguide - Success Rate | Without Endoguide
Number analyzed (Participants) | 555 | 449
participants | 555 | 449

2. Secondary Outcome: Perception of Pain
Description: VAS (Visual Analogue Scale), 0 - 10. VAS 0 is no pain, VAS 10 is max pain. Scores on a scale
Time Frame: After endoscopy (within 10mins) and 1 day after endoscopy
Measure: Mean (Standard Deviation); unit: Scores on a scale 0-10
Arm/Group | With Endoguide | Without Endoguide
Number analyzed (Participants) | 555 | 449
Scores on a scale 0-10
  Score within 10mins of endoscopy | 3.84 (2.78) | 4.12 (2.98)
  Score 1 day after endoscopy | 3.56 (2.90) | 3.72 (3.15)

ADVERSE EVENTS:
Arm/Group | With Endoguide | Without Endoguide
Serious Adverse Events (participants affected / at risk) | 0/555 | 0/449
Other Adverse Events (participants affected / at risk) | 0/555 | 0/449

LIMITATIONS AND CAVEATS:
Early termination due to higher than expected eligible patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes